CLINICAL TRIAL: NCT04236375
Title: The Development of an Artificial Intelligence Platform for Screening and Referral of Cognitive Dysfunction
Brief Title: Eye Movement and Cognitive Dysfunction
Acronym: EMCD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Professor, Sun Yat-sen University
Other Study IDs: Eye movement-cognitive decline
Record Dates: First submitted 2020-01-18; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Eye Movement Disorder; Cognitive Dysfunction
MeSH Terms: conditions — Ocular Motility Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Normal: Subjects over 45 years old without cognitive dysfunction
- Mild cognitive decline: Subjects who are diagnosed as mild cognitive decline(MCI) according to neurologists.
- Alzheimer's disease: Subjects who are diagnosed as Alzheimer's disease(AD) according to neurologists.
- Vascular dementia: Subjects who are diagnosed as vascular dementia(VD) according to neurologists.
- Lewy body dementia: Subjects who are diagnosed as Lewy body demenita (DLB) according to neurologists.
- Frontotemporal dementia: Subjects who are diagnosed as Frontotemporal demenita (FD) according to neurologists.
- Other dementia: Subjects who are diagnosed as dementia but are not as AD, VD, DLB OR FD.

SUMMARY:
There is association between eye movement disorder and cognitive dysfunction. Therefore, utilizing eye movement and screening for cognitive dysfunction is feasible. In the present study, we will develop an artificial intelligence platform to screening for cognitive dysfunction by inspecting the function of eye movement. Futher more, based on the screening results, the platform will offer referral suggestions.

ELIGIBILITY:
Inclusion Criteria:

* ①Subjects who are diagnosed as mild cognitive decline, Alzheimer's disease, Vascular dementia, Lewy body dementia, Frontotemporal dementia, other dementia and normal by neurologist.
* ②Subjects who can cooperate with the inspection.
* ③Subjects who agree to participate in the study and sign the consent form

Exclusion Criteria:

* ①Subjects who cannot do the inspection.
* ②Subjects who suffer from diseases that compromise the inspection.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who are over 45 years old with or without cognitive dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Area under the curve | up to 1 month
  AUC values for predicting whether subject has cognitive impairment or not

SECONDARY OUTCOMES:
Accuracy, true positive rate, and true negetive rate | up to 1 month
  The performance of this artificial platform

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D.,Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Xun Wang, M.D.,Ph.D, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Shuyi Zhang, M.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University